CLINICAL TRIAL: NCT00629161
Title: Clinical Trial on the Effectiveness of Traditional Chinese Medicinal Mixture in Parkinson Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Dingfang Cai, Zhongshan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006BAI04A11-3
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental)
  Interventions: Drug: Traditional Chinese Medicinal Mixture (composed of Roucongrong and adjuvant)
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Traditional Chinese Medicinal Mixture (composed of Roucongrong and adjuvant) — 12 months period of Traditional Chinese Medicinal Mixture per day plus 1 month wash-out period without herbal medicine
  Arms: A
Drug: placebo — 12 months period of placebo plus 1 month period without placebo
  Arms: B

SUMMARY:
This study was designed to evaluate the symptomatic effects or potential disease progression slowing down effect of a kind of Traditional Chinese Medicinal Mixture in Parkinson's disease (PD) patients. The treatment phase includes 12 months period of Traditional Chinese Medicinal Mixture per day or placebo and 1 month wash-out period without herbal medicine and placebo.

DETAILED DESCRIPTION:
The design of the study was a prospective, randomized, multicenter, double-blind placebo-controlled protocol. The intervention includes Traditional Chinese Medicinal Mixture tid or matched placebo.

Participating study centers include Neurological University Outpatient Clinics and Neurological Departments of Community-based Hospitals experienced with PD patients.

The primary outcome measure was the combined Unified Parkinson's Disease Rating Scale (UPDRS).

The hypothesis of this study was that Traditional Chinese Medicinal Mixture improves the overall wellbeing of PD patients and thus may leads to an improvement of parkinsonian symptoms in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease according to the UK Brain Bank criteria
* Hoehn & Yahr stadium Ⅰ～Ⅲ
* Age over 50 years
* Taking only levodopa and/or dopamine agonists when recruiting
* Consistent with the liver kidney deficiency type by Traditional Chinese Medicine (TCM) standard
* Patients voluntarily take part in this study and signed the informed consent

Exclusion Criteria:

* Modified Hoehn-Yahr scale are higher than 4
* Had other serious illness such as liver/kidney failure, serious infection etc
* Allergic to the study drug
* Had been participated in other clinical trials during the last 3 months prior to study inclusion.
* Taking Coenzyme Q10, MAO-B inhibitors, or vitamin E, all of which might improve the symptom or slowdown the progression of PD.
* Taking herbal medicine that can nourish the liver and kidney by TCM standard.
* Had serious mental disorder and could not describe his/her symptom.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | 13 months

SECONDARY OUTCOMES:
Hoehn & Yahr scale | 13 months
Schwab & England score | 13 months
The liver kidney deficiency scale score by Traditional Chinese Medicine standard | 13 months
Dose of levodopa per day | 13 months
Dose of dopamine Agonists per day | 13 months
Parkinson disease sleep scale (PDSS) | 13 months
Assessment of autonomic dysfunction in Parkinson disease (SCOPA-AUT) | 13 months
Changes in laboratory indexes as safety assessment, including red blood cell(RBC), white blood cell(WBC), platelet(PLT), alanine transaminase(ALT), aspartate transaminase (AST), blood urea nitrogen (BUN), creatinine(Cr) in blood samples, ect. | 12 months

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Department of Neurology, Xuanwu hospital, Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Department of Neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Nuerology, Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanghai Chinese Medical Hospital, Shanghai, Shanghai Municipality
  - Department of Nuerology, Xinhua Hospital, Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The Sixth People's Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Department of Neurology, Yueyang Hospital of Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Department of Neurology, The second people's hospital of Wenzhou, Wenzhou, Zhejiang